# **Teaching Academic Success Skills to Students with Autism Spectrum Disorders in the Clinical Setting**

Study Protocol and Statistical Analysis Plan

Clinical Trials.gov Identifier: NCT03606343

**September 22, 2020** 

# **STUDY PROTOCOL**

## **PURPOSE OF STUDY:**

The goal of the study is to develop an academic EF intervention, *Achieving/Academic Independence in Middle School (AIMS)*, for high functioning (i.e., IQ score ≥80) middle-school youth with ASD and EF deficits. The primary aim is to: Examine the feasibility and acceptability of AIMS in a series of open trials (n=21) including the feasibility of: 1) implementing the measurement protocol, 2) operationalizing intervention delivery, 3) assessing both trained and untrained areas of functioning, 4) assessing whether improvements in academic EF skills (*proposed mechanism of treatment*) are related to functional educational outcomes (e.g., homework behaviors, grades), and 5) exploring the data for potential treatment moderators (e.g., gender, severity). It is hypothesized that AIMS will be feasible, acceptable (attendance, satisfaction), and will result in improved academic EF skills associated with reduced academic impairment and homework problems.

### **STUDY DESIGN:**

Open Trial: To document proof of concept and gather sufficient preliminary data for a future RCT, 3 cohorts of youth with ASD (n=21) will be recruited (three groups will be recruited to participate in the group intervention; the maximum group size for this intervention is 7 based on the level of individualized attention needed during the intervention). A research assistant will observe all sessions and complete treatment fidelity checklists to monitor adherence. Sessions will also be videotaped for later use (e.g., training, fidelity coding). The primary teacher will complete organization and time management checklists weekly. We do not anticipate making major changes to the intervention during the open trials; however, as needed the intervention manual may be refined to be clearer. Parent(s) and their teen will attend 7 intervention sessions offered 1 week apart at CCHMC. Session content will include psychoeducation about the academic EFs in ASD and will be taught strategies and skills targeting these deficits, including using a behavioral contract (i.e., Agreement), organization skills (e.g., homework system, binder organization, etc.), time management skills (e.g., planner), problem solving skills, and study skills (e.g., flash cards). We will also be doing midweek check-ins with parents during the intervention to increase accountability and coach parents as needed.

Post Assessment and Exit Interviews: The primary measures collected will be treatment fidelity and academic EF skills acquisition, although other measures will be collected to pilot these measures and methods for collection and to gather information about whether they capture gains made by families. Parents and youth with ASD will also be surveyed regarding their experience of the intervention and whether they understood intervention materials in exit interviews.

Consultation with Experts: A webinar will be scheduled to process the information obtained during the open trial, including the feedback from the parents, and youth obtained in the exit interviews, the fidelity ratings, the utility and feasibility of the proposed measures.

Finalize Intervention Manual: A finalized draft of the manual will be developed including sections on troubleshooting, treatment rationale, strategies for specific skills, case examples, and

guidance for establishing and maintaining effective relationships with participants<sup>68</sup> will be incorporated. Finalized graphics and storyboards will be selected and scripts revised for the animated clips depicting important content.

## **Participants**

Youth with ASD: The target population is high functioning middle school youth (6, 7, and 8<sup>th</sup> graders ages 10 to 14) who have an educational label of Autism (e.g., school referred) and/or meet diagnostic criteria for ASD (e.g., clinic referred). In cases where it may need to be clarified (e.g., youth attends a specialized school for ASD, or the child is in an intermediate school), we will confirm that youth transition between teachers for core academic subjects. For research purposes, the diagnosis of all youth will be confirmed using the ADOS-2. All participants with ASD will present with EF problems based on the parent or teacher rated BRIEF-2 T-Score >60 on the Planning, Organization, or Monitor subscales.

An IQ score  $\geq$ 80 will be required in order to select a high functioning population that will be most likely to profit from the intervention and are more likely to be in the mainstreamed educational environment or be eligible for mainstreaming.

Youth in middle school (typical age range 10 to 14) attending public or private middle/junior high schools will be recruited. Youth receiving pullout special education services for the majority of the day will be excluded because services required for those individuals would exceed that which AIMS could address. Additionally, those who receive significant support in the classroom (e.g., one-on-one aide for the whole school day) may not benefit from the intervention given its focus on promoting independence and initiative; this will be verified by reviewing the IEP.

Both sexes will be represented although more males than females (4:1 ratio) are anticipated given prevalence data for ASD<sup>69</sup>.

Parents/Caregivers of Youth with ASD: Since parents/caregivers will be critically involved in implementing and reinforcing the intervention components, their input will be invaluable. Parents will be the primary caregiver of a child with high functioning ASD, English-speaking, and be willing and able to attend the intervention sessions.

*Expert Consultants:* An expert panel of consultants with expertise in academic issues facing youth with ASD and with developing and implementing school-based interventions will provide feedback on the final manual.

<u>Measures</u>: Measures collected will include information on family background, and measures assessing eligibility, EF, academic functioning, self-determination, parent-child relationship and satisfaction. Also see Table 1.

### Participant Demographics & Eligibility:

Family Demographic/Developmental History: Includes family status, parent occupation, education, medical and developmental history, school history (including special education placements) completed by parents.

Autism Diagnostic Observation Schedule, 2<sup>nd</sup> Edition (ADOS-2)<sup>70</sup> is the "gold standard" clinician-administered assessment that will examine social interaction, language and communication, and restricted and repetitive behaviors and interests. All youth will be administered Module 3 of the ADOS-2 to confirm ASD diagnosis. Note that if an ADOS-2 has

been administered within the past two years by staff at CCHMC, parents will be asked to sign a release of information form and the results from that assessment will be obtained.

Kaufman Brief Intelligence Tests-2 (K-BIT)<sup>71</sup>: The K-BIT is a culturally-sensitive standardized assessment that estimates verbal and non-verbal and overall intelligence. This test has good reliability and validity and will be administered to confirm that the participant has an  $IQ \ge 80$ . Note that if a K-BIT has been administered within the past year for other research studies at CCHMC, parents will be asked to sign a release of information form and the results from that assessment will be obtained.

## **Executive Functioning**

Behavior Rating Inventory of Executive Function (BRIEF)<sup>73</sup>: Parents and teachers will complete the BRIEF assessing EF behaviors in the home and school environments.

Children's Organizational Skills Scale (COSS)<sup>74</sup>: Parents, teens, and teachers will complete the COSS assessing multiple facets of a child's organizational skills.

## **Academic Functioning**

Subtests of the Woodcock Johnson Tests of Achievement III (WJ)<sup>76</sup>: Reading Comprehension (#9,#17), Basic Writing Cluster (#7,# 16), Math Reasoning Cluster (#10, #18), and the Academic Knowledge subtest (# 19) will be administered to assess academic achievement in student participants.

Homework Problems Checklist (HPC)<sup>77</sup>: The HPC is a parent-report instrument that is commonly used as a screening tool for and outcome measure of homework problems.

Classroom Performance Survey (CPS)<sup>78</sup>: The CPS, completed by teachers, is a measure of academic impairment specifically designed for secondary school youth. A shorter variant of this scale will be completed by teachers on a weekly basis while the child is attending the intervention.

Academic Performance Rating Scale (APRS)<sup>79</sup>: The APRS is a 19-item scale that is completed by the teacher that measures how well the child is performing academically in the classroom.

#### Parent-Youth Relationship

Parenting Relationship Questionnaire (PRQ)<sup>80</sup>. The PRQ is a parent-report instrument reporting on how parents feel about their children and the task of parenting. Subscales include Communication, Involvement, Satisfaction with School, Parenting Confidence, Relational Frustration, Attachment, and Discipline Practices. Lower T-scores indicate greater severity of relationship problems. This measure is included to assess whether parents report improvements in communication, satisfaction with school, increased confidence, and decreased frustration.

| Table 1. Measures | Rater | Time | Eligibility | Pre | AIMS | Post | Domain |
|---|---|---|---|---|---|---|---|
| Autism Diagnostic Observation Schedule | Y | 60 | X | | | | |
| Kaufman Brief Intelligence Test – Second Ed. (KBIT-2) | Y | 20 | X | | | | |
| Behavior Rating Inventory of Executive Function Second<br>Edition (BRIEF-2) | P, T | 10 | X | | | X | EF |
| Children's Organizational Skills Scale (COSS) | P,<br>T,Y | 10 | | X | | X | EF |
| Woodcock Johnson (WJ-IIII) Achievement Subtests | Y | 30 | | X | | X | A |
| Homework Problems Checklist (HPC) | P | 5 | | X | | X | A |
| Classroom Performance Survey (CPS) | T | 10 | | X | | X | A |
| Academic Performance Rating System (APRS) | T | 10 | | X | | X | A |

| Parenting Relationship Questionnaire (PRQ) | P | 10- | X | X | PY |
|--------------------------------------------|---|-----|---|---|----|
| | | 15 | | | |

Y = Youth, P = Parent, T = Teacher, EF = academic executive functioning skill, A = academic outcome, PY=Parent-Youth relationship, I = Independence/Initiative, S = Satisfaction

## **Recruitment and Informed Consent**

The investigative team has considerable experiencing with recruiting and retaining youth with ASD in intervention studies and recruitment difficulties are not anticipated. The team has well-established contacts with public and private school systems in Cincinnati and surrounding areas, and notices will be placed in schools to alert teachers and parents about this research opportunity. Clinicians and physicians at the Kelly O'Leary Center (TKOC) for Autism, the Division of Developmental Behavioral Pediatrics, and the Division of Psychiatry at Cincinnati Children's Hospital Medical Center's (CCHMC) will also be notified about this opportunity. Participants with ASD will also be recruited from local schools, including those specializing in ASD, as well as from the TKOC.

At <u>TKOC</u>, students will be identified through a variety of resources including (1) an existing database of children and adolescents who were previously assessed and diagnosed with an ASD at TKOC; (2) Dr. Duncan's existing research database of 150 youth with ASD who have participated in her previous studies; (3) an existing research database of ~60 youth with ASD who have participated in studies through the CCHMC Psychiatry Department; (4) treatment referrals from clinicians at TKOC and community providers. Currently, there are 178 youth between the ages of 10 to 14 years, which is the typical age of middle schoolers, who were evaluated or received treatment at TKOC in 2017 and could be recruited for the current research study; additionally, there are 94 individuals in this age range on the waitlist for services at TKOC that could also be approached. Families may be sent a letter indicating that they were identified because of having been seen previously at TKOC along with a "do not contact" postcard. Families not returning the postcards will be called by research staff to share more about the study and invite participation.

At <u>schools</u>, Student Services Directors, Special Educators, school mental health professionals, and/or teachers will be approached to identify high functioning middle school students with ASD who might be interested in participating. These individuals will be provided with a recruitment letter and flyer to distribute to parents of these youth. Students with an Individualized Education Program (IEP) that includes items related to EF (e.g., organization challenges), or whom teachers and/or school MHPs consider as having significant challenges in these domains will be of particular interest.

Participants may be recruited using IRB-approved materials including advertising and/or print, electronic, social and digital media, news/broadcast, face-to-face marketing and flyers at Cincinnati Children's and in the community. Some of these recruitment materials will direct potential participants to a REDCap e-screener page where potential participants will be directed to provide contact information so that study staff may contact the participants to inform them about the study.

An initial eligibility screen will be conducted by telephone which will include asking parents to give verbal permission for us to contact the teacher to complete the BRIEF-2. Eligible families will be invited to an in-person screening visit at CCHMC. At the in person screening visit, the consent form and assent form, which are written in a language that is understandable to parents and teens, will be reviewed in detail. The consent form will also clarify that their data will be shared with other researchers via the National Database for Autism Research (NDAR) without exposing personally identifiable information. Upon conclusion of the review, the project

coordinator will ask if the parent and child are still interested in the study and if they are willing to sign the consent/assent forms— one will be provided for the family to keep for their records and one to sign for the study. We may consent the families electronically and send them an electronic copy of the consent/assent forms via REDCap. After signing the consent/assent forms, the baseline assessment battery will commence. This will include the a) ADOS-2<sup>70</sup> to assess ASD symptoms, the Stanford-Binet 5<sup>th</sup> Edition<sup>72</sup> to confirm IQ, and the BRIEF-2 to confirm EF difficulties. For those youth who meet criteria, additional measures will be administered either at the screening visit or at a second visit depending on the families' wishes and fatigue level, assessing the outcomes of interest (e.g., Homework Problems Checklist, academic testing). We will also be asking the parents to bring a copy of their child's school IEP in order to determine if they fit criteria of being in a mainstream classroom for majority of the day without too much support from school staff.

Teachers are also participants in this study as they complete ratings of academic functioning that are critical to the study aims. Thus, engaging and retaining school personnel throughout the study will be important. The PIs will provide an overview of the study to teachers and provide an opportunity to ask questions as needed. The importance of teacher participation will be emphasized as crucial to accomplishing the aims of the study. In addition, teachers will be compensated for their time and effort in completing ratings.

# **STATISTICAL ANALYSIS PLAN**

Descriptive statistics will summarize attendance, satisfaction (AIQ), fidelity, drop-out rates, exit interview data to assess feasibility and acceptability. Within group (pre-test, post-test) mixed factorial ANCOVAs controlling for pre-test scores will test for the presence of improvements. It is hypothesized that youth with ASD will demonstrate improved academic EF skills (BRIEF-2, COSS, HPC). The primary analytic focus will be on evaluating whether the observed effect sizes across outcomes warrant continued study of AIMS as a treatment strategy. A moderate (i.e., Cohen's  $d = .5^{81}$ ) effect size for academic EF measures will be evidence of significant improvement. We will explore whether AIMS improves academic (WJ, CPS, APRS), and parent-child relationship (PRQ) outcomes between pre- and post- assessments. Correlations between changes in academic EF skills and changes in the other outcomes measures will also be computed to explore whether changes in academic EF skills are related to functional academic outcomes, as these are the primary target and proposed mechanism of treatment.

<u>Exploratory Analyses</u>: We will also explore potential moderators such as sex, IQ, ASD and EF severity, and socioeconomic status qualitatively and with non-parametric statistics given the lack of power.

### References

- 1. Whitby PJS, Mancil GR. Academic achievement profiles of children with high functioning autism and asperger syndrome: A review of the literature. *Education and Training in Developmental Disabilities*. 2009;44(4):551-560.
- 2. Nation K, Clarke P, Marshall CM, Durand M. Hidden language impairments in children: parallels between poor reading comprehension and specific language impairment? *J Speech Lang Hear Res.* 2004;47(1):199-211.
- 3. Wagner M, Marder C, Blackorby J, et al. *The achievements of youth with disabilities during secondary school: A report from the National Longitudinal Transition Study-2*. Menlo Park2003.
- 4. Keen D, Webster A, Ridley G. How well are children with autism spectrum disorder doing academically at school? An overview of the literature. *Autism.* 2016;20(3):276-294.
- 5. Ashburner J, Ziviani J, Rodger S. Surviving in the mainstream: Capacity of children with autism spectrum disorders to perform academically and regulate their emotions and behavior at school. *Research in autism spectrum disorders*. 2010;4(1):18-27.
- 6. Wolf LE, Thierfeld Brown J, Kukiela GR. *Students with Asperger Syndrome: A Guide for College Personnel*. Shawnee Mission: Autism Asperger Publishing Co.; 2009.
- 7. Jones CR, Happe F, Golden H, et al. Reading and arithmetic in adolescents with autism spectrum disorders: peaks and dips in attainment. *Neuropsychology*. 2009;23(6):718-728.
- 8. Troyb E, Orinstein A, Tyson K, et al. Academic abilities in children and adolescents with a history of autism spectrum disorders who have achieved optimal outcomes. *Autism*. 2014;18(3):233-243.
- 9. Endedijk H, Denessen E, Hendriks AW. Relationships between executive functioning and homework difficulties in students with and without autism spectrum disorder: An analysis of student- and parent-reports. *Learn Ind Diff.* 2011;21:765–770.
- 10. Hampshire PK, Butera GD, Dustin TJ. Promoting Homework Independence for Students With Autism Spectrum Disorders. *Int School Clin.* 2014;49(5):290-297.
- 11. Best JR, Miller PH, Naglieri JA. Relations between executive function and academic achievement from ages 5 to 17 in a large, representative national sample. *Learn Ind Diff.* 2011;21(4):327-336.
- 12. Best JR, Miller PH, Jones LL. Executive functions after age 5: Changes and correlates. *Dev Rev.* 2009;29(3):180-200.
- 13. Fisher N, Happe F. A training study in theory of mind and executive function in children with autistic spectrum disorders. *J Autism Dev Disord*. 2005;35:757–771.
- 14. Gioia GA, Isquith PK, Kenworthy L, Barton RM. Profiles of everyday executive function in acquired and developmental disorders. *Child Neuropsychol.* 2002;8:121-137.
- 15. Blijd-Hoogewys EM, Bezemer ML, van Geert PL. Executive functioning in children with ASD: an analysis of the BRIEF. *J Autism Dev Disord*. 2014;44(12):3089-3100.
- 16. Kenworthy L, Black DO, Wallace GL, Ahluvalia T, Wagner AE, Sirian LM. Disorganization: the forgotten executive dysfunction in high-functioning autism (HFA) spectrum disorders. *Dev Neuropsychol.* 2005;28(3):809-827.
- 17. Pennington BF, Ozonoff S. Executive functions and developmental psychopathology. *J Child Psychol Psychiatry*. 1996;37(1):51-87.
- 18. Hill EL. Executive dysfunction in autism. *Trends Cogn Sci.* 2004;8(1):26-32.

- 19. Hill EL, Bird CM. Executive processes in Asperger syndrome: patterns of performance in a multiple case series. *Neuropsychologia*. 2006;44(14):2822-2835.
- 20. Fleury VP, Hedges S, Hume K, et al. Addressing the academic needs of adolescents with Autism Spectrum Disorder in secondary education. *Rem Spec Educ.* 2014;35(2):68-79.
- 21. Ruble LA, Scott MM. Executive functions and the natural habitat behaviors of children with autism. *Autism.* 2002;6(4):365-381.
- 22. Rogers SJ. Neuropsychology of Austim in young children and its implications for early intervention. *Ment Retard Dev Disabil Res Rev.* 1998;4:104-112.
- 23. Myles BS, Simpson RL. Asperger Syndrome: An Overview of Characteristics. *Focus on Autism and Other Developmental Disabilities*. 2002;17:132-137.
- 24. Janeslatt G, Granlund M, Kottorp A. Measurement of time processing ability and daily time management in children with disabilities. *Disability and health journal*. 2009;2(1):15-19.
- 25. Clark CA, Pritchard VE, Woodward LJ. Preschool executive functioning abilities predict early mathematics achievement. *Dev Psychol.* 2010;46(5):1176-1191.
- 26. Wallace GL, Kenworthy L, Pugliese CE, et al. Real-world executive functions in adults with Autism Spectrum Disorder: Profiles of impairment and associations with adaptive functioning and co-morbid anxiety and depression. *J Autism Dev Disord*. 2016;46(3):1071-1083.
- 27. McEvoy RE, Rogers SJ, Pennington BF. Executive function and social communication deficits in young autistic children. *J Child Psychol Psychiatry*. 1993;34(4):563-578.
- 28. Gokcen E, Frederickson N, Petrides KV. Theory of Mind and Executive Control Deficits in Typically Developing Adults and Adolescents with High Levels of Autism Traits. *J Autism Dev Disord*. 2016;46(6):2072-2087.
- 29. Leung RC, Vogan VM, Powell TL, Anagnostou E, Taylor MJ. The role of executive functions in social impairment in Autism Spectrum Disorder. *Child Neuropsychol*. 2016;22(3):336-344.
- 30. DuPaul GJ, Stoner G. *ADHD in the schools: Assessment and intervention strategies.* 2 ed. New York: Guilford Press; 2003.
- 31. Goldstein G, Minshew NJ, Siegel DJ. Age differences in academic achievement in high-functioning autistic individuals. *J Clin Exp Neuropsychol*. 1994;16(5):671-680.
- 32. Adreon D, Stella J. Transition to middle and high School: Increasing the success of students with Asperger Syndrome. *Int School Clin.* 2001;36(5):268-271.
- 33. Mullins ER, Irvin JL. Transition into middle school: What research says. *Middle School Journal*. 2000;31(3):57-60.
- 34. Whitby PJS. The Effects of "Solve It!" on the Mathematical Word Problem Solving Ability of Adolescents with Autism Spectrum Disorders. *Focus on Autism and Other Developmental Disabilities*. 2013;28(2):78-88.
- 35. Eccles JS. Schools, academic motivation, and stage-environment fit. In: Lerner RM, Steinberg LD, eds. *Handbook of adolescent psychology*. 2 ed. New York: Wiley; 2004:125–153.
- 36. Evans SW, Axelrod J, Langberg JM. Efficacy of a school-based treatment program for middle school youth with ADHD: pilot data. *Behav Modif.* 2004;28(4):528-547.
- 37. Evans SW, Langberg J, Raggi V, Allen J, Buvinger EC. Development of a school-based treatment program for middle school youth with ADHD. *J Atten Disord*. 2005;9(1):343-353.

- 38. Abikoff HA, Gallagher R, Wells KC, et al. Remediating organizational functioning in children with ADHD: Immediate and long-term effects from a randomized controlled trial. *J Consult Clin Psychol*. 2013;81(1):113-128.
- 39. Tamm L, Vaughn A, Leavitt M, et al. Academic success groups for adolescents with ADHD. Paper presented at: Biennial Meeting of the Society for Research in Child Development2015; Philadelphia, PA.
- 40. Langberg JM, Epstein JN, Girio EL, Becker SP, Vaughn AJ, Altaye M. Materials Organization, Planning, and Homework Completion in Middle School Students with ADHD: Impact on Academic Performance. *School Ment Health*. 2011;3(2):93-101.
- 41. Abikoff HA, Gallagher R. Assessment and remediation of organizational skills deficits in children with ADHD. In: McBurnett K, Pfiffner L, eds. *Attention Deficit Hyperactivity Disorder: Concepts, controversies, new directions*. New York: Information Healthcare; 2008:137–152.
- 42. Ciesielski HA, Tamm L, Vaughn A, Cyran J, Epstein JN. Academic success groups for middle-school children with ADHD in the outpatient mental health setting. *J Atten Disord*. in press.
- 43. Vaughn AJ, Tamm. L, Loren R, Ciesielski H, Cyran J. Academic Success Groups for Middle School Children with ADHD. Paper presented at: 48th Annual Association of Behavioral and Cognitive Therapy (ABCT)2014; Philadelphia, PA.
- 44. Langberg JM. *Improving children's homework, organization, and planning skills: A parent's guide.* Bethesda: National Association of School Psychologists; 2014.
- 45. Courchesne E, Pierce K. Brain overgrowth in autism during a critical time in development: implications for frontal pyramidal neuron and interneuron development and connectivity. *Int J Dev Neurosci.* 2005;23(2-3):153-170.
- 46. Bearss K, Lecavalier L, Minshawi N, et al. Toward an exportable parent training program for disruptive behaviors in autism spectrum disorders. *Neuropsychiatry (London)*. 2013;3(2):169-180.
- 47. Ingersoll B, Dvortcsak A. Including parent training in the early childhood special education curriculum for children with Autism Spectrum Disorders. *J Pos Behav Int.* 2006;8(2):79-87.
- 48. Chiang HM, Cheung YK, Li H, Tsai LY. Factors associated with participation in employment for high school leavers with autism. *J Autism Dev Disord*. 2013;43(8):1832-1842.
- 49. Doren B. The relationship between parent expectations and postschool outcomes of adolescents with disabilities. *Exceptional children*. 2012;79:7-23.
- 50. Kirby AV. Parent Expectations Mediate Outcomes for Young Adults with Autism Spectrum Disorder. *J Autism Dev Disord*. 2016;46(5):1643-1655.
- 51. McDonald TA, Machalicek W. Systematic review of intervention research with adolescents with autism spectrum disorders. *Research in autism spectrum disorders*. 2013;7(11):1439-1460.
- 52. Dorminy KP, Luscre D, Gast DL. Teaching Organizational Skills to Children with High Functioning Autism and Asperger's Syndrome. *Education and Training in Developmental Disabilities*. 2009;44(4):538 –550.
- 53. Brown KE, Mirenda P. Contingency mapping: Use of a novel visual support strategy as an adjunct to functional equivalence training. *J Pos Behav Int.* 2006;8(3):155-164.
- 54. Wilczynski SM, Fusilier I, Dubard M, Elliott A. Experimental analysis of proximity as a

- social stimulus: Increasing on-task behavior of an adolescent with autism. *Psychology in the Schools*. 2005;42(2):189-196.
- 55. Kenworthy L, Anthony LG, Naiman DQ, et al. Randomized controlled effectiveness trial of executive function intervention for children on the autism spectrum. *J Child Psychol Psychiatry*. 2014;55(4):374-383.
- 56. Wilkinson LA. Autism spectrum disorder in children and adolescents: Evidence-based assessment and intervention in schools. Washington, DC, US: American Psychological Association; 2014.
- 57. Keehn RHM, Lincoln AJ, Brown MZ, Chavira DA. The Coping Cat program for children with anxiety and autism spectrum disorder: A pilot randomized controlled trial. *J Autism Dev Disord*. 2013;43:57-67.
- 58. White SW, Albano AM, Johnson CR, et al. Development of a cognitive-behavioral intervention program to treat anxiety and social deficits in teens with high-functioning autism. *Clin Child Fam Psychol Rev.* 2010;13(1):77-90.
- 59. <a href="http://depts.washington.edu/camp2013/Apex Summer Camp/About.html">http://depts.washington.edu/camp2013/Apex Summer Camp/About.html</a>.
- 60. Robin AL, Foster SL. Negotiating parent-adolescent conflict: A behavioral-family systems approach. New York: The Guilford Press; 1989.
- 61. Field S, Hoffman A. The importance of family involvement for promoting self-determination in adolescents with autism and other developmental disabilities. *Focus on Autism and Other Developmental Disabilities*. 1999;14(1):36-41.
- 62. Carter EW, Lane KL, Cooney M, Weir K, Moss CK, Machalicek W. Parent assessments of self-determination importance and performance for students with autism or intellectual disability. *Am J Intellect Dev Disabil*. 2013;118(1):16-31.
- 63. Lee SH, Simpson RL, Shogren KA. Effects and implications of self-management for students with Autism: A meta-analysis *Focus on Autism and Other Developmental Disabilities*. 2007;22(1):2-13.
- 64. Hume K, Loftin R, Lantz J. Increasing independence in autism spectrum disorders: a review of three focused interventions. *J Autism Dev Disord*. 2009;39(9):1329-1338.
- 65. Olympia DE, Sheridan SM, Jenson W. Homework: A Natural Means of Home-School Collaboration. *School Psychol Quart*. 1994;9(1):60-80.
- 66. Cooper H, Robinson JC, Patall EA. Does homework improve academic achievement? A synthesis of research, 1987–2003. *Review of Educational Research*. 2006;76(1):1-62.
- 67. Epstein JL. *Homework practices, achievements, and behaviors of elementary school students*. Baltimore: Center of Research on Elementary and Middle schools, Johns Hopkins University;1988. 26.
- 68. Carroll KM, Nuro KF. One size cannot fit all: A stage model for psychotherapy manual development. *Clin Psychol Sci Prac*. 2002;9(4):396-406.
- 69. American Psychiatric Association. *Diagnostic and Statistical Manual of Mental Disorders*. 5 ed. Washington D.C.: Author; 2013.
- 70. Lord C, Rutter M, DiLavore PC, Risi S, Gotham K, Bishop SL. *Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) Modules 1-4*. Los Angeles, California: Western Psychological Services; 2012.
- 71. Kaufman AS, Kaufman NL. *Kaufman Brief Intelligence Test Second Edition*. Circle Pines: AGS; 2004.
- 72. Roid GH. Stanford-Binet Intelligence Scales 5th ed: Riverside Publishing; 2003.
- 73. Gioia GA, Isquith PK, Guy SC, Kenworthy L. Behavior Rating Inventory of Executive

- Function Professional Manual. Lutz: Psychological Assessment Resources, Inc; 2000.
- 74. Abikoff HA, Gallagher R. *The Children's Organizational Skills Scales Technical Manual*. North Tonawanda: Multihealth Systems, Inc; 2009.
- 75. Langberg JM, Smith BH. Developing evidence-based interventions for deployment into school settings: A case example highlighting key issues of efficacy and effectiveness. *Eval Program Plann.* 2006;29(4):323-334.
- 76. Woodcock RW, McGrew KS, Mather N. Woodcock-Johnson III. Itasca: Riverside; 2001.
- 77. Anesko KM, Schoiock G, Ramirez R, Levine FM. The Homework Problem Checklist: Assessing children's homework problems. *Behavioral Assessment*. 1987;9:179–185.
- 78. Brady CE, Evans SW, Berlin KS, Bunford N, Kern L. Evaluating school impairment with adolescents using the classroom performance survey. *School Psychol Rev.* 2012;41(4):429-446.
- 79. DuPaul GJ, Rapport MD, Perriello LM. Teacher ratings of academic skills: The development of the Academic Performance Rating Scale. *School Psychol Rev.* 1991;20:284-300.
- 80. Kamphaus RW, Reynolds CR. *Parenting Relationship Questionnaire*. Minneapolis: Sage Publications, Inc; 2006.
- 81. Cohen J. Statistical Power Analysis for the Behavioral Sciences Second Edition. Hillsdale: Lawrence Erlbaum Associates; 1988.
- 82. Becker SP. *Child Concentration Inventory, Second Edition (CCI-2).* Cincinnati, OH: Author; 2015.
- 83. Sáez B, Servera M, Burns GL, Becker SP. Validity of children's self-report of sluggish cognitive tempo: Correspondence with parent and teacher measure. *Under review.* 2018.
- 84. Becker SP, Leopold DR, Burns GL, et al. The internal, external, and diagnostic validity of sluggish cognitive tempo: A meta-analysis and critical review. *Journal of the American Academy of Child and Adolescent Psychiatry*. 2016;55(3):163-178.
- 85. Burns GL, Lee S, Servera M, McBurnett K, Becker SP. *Child and Adolescent Behavior Inventory Parent Version 1.0.* Pullman, WA: Author; 2015.
- 86. Burns GL, Lee S, Servera M, McBurnett K, Becker SP. *Child and Adolescent Behavior Inventory Teacher Version 1.0.* Pullman, WA: Author; 2015.
- 87. Sáez B, Servera M, Becker SP, Burns GL. Optimal items for assessing sluggish cognitive tempo in children across mother, father, and teacher ratings. *Journal of Clinical Child and Adolescent Psychology*. 2018.
- 88. Becker SP, Burns GL, Schmitt AP, Epstein JN, Tamm L. Toward establishing a standard symptom set for assessing sluggish cognitive tempo in children: Evidence from teacher ratings in a community sample. *Assessment*. 2017.